CLINICAL TRIAL: NCT04111133
Title: Efficacy of Carvedilol + Ivabradine vs Carvedilol Alone for Left Ventricular Diastolic Dysfunction in Chronic Liver Disease Patients and Its' Impact on Morbidity and Mortality; a Prospective Randomized Controlled Trial.
Brief Title: Ivabradine in Cirrhotic Cardiomyopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant Professor and Principal Investigator, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2019/001617
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Cirrhotic Cardiomyopathy; Left Ventricular Dysfunction; Cirrhosis, Liver; Portal Hypertension
Keywords: Cirrhotic cardiomyopathy; Left ventricular diatolic dysfunction; Carvedilol; Ivabradine
MeSH Terms: conditions — Ventricular Dysfunction, Left; Liver Cirrhosis; Hypertension, Portal | interventions — Ivabradine

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carvedilol + Ivabradine (Experimental)
  Interventions: Drug: Betablocker + ivabradine
- Carvedilol (Active Comparator)
  Interventions: Drug: Betablocker

INTERVENTIONS:
Drug: Betablocker + ivabradine — Use of maximum tolerated dose of carvedilol and ivabradine to achieve therapeutic heart rate reduction (THR) to 55-65 beats per minute
  Arms: Carvedilol + Ivabradine
Drug: Betablocker — Use of maximum tolerated dose of carvedilol to achieve targeted heart rate reduction (THR) to 55-65 beats per minute (responder) or inability to reach THR (non responder) with maximum dose of carvedilol, maintaining a minimum MAP of 70 mmHg.
  Arms: Carvedilol

SUMMARY:
A total of 130 patients with liver cirrhosis who fulfill the criteria of the study, and who have been found to have left ventricular diastolic dysfunction on a screening 2D echocardiography, will then be randomized by Block randomization technique, to two arms in a ratio 1:1(Group A) will receive carvedilol+ Ivabradine targeted therapy for heart rate reduction while Group B will receive Carvedilol alone; and the dosage of drug in the treatment arm will be titrated every week to achieve target heart rate of 50-60/ minute. Patients in the treatment arms, who are unable to tolerate carvedilol due to hypotension episodes, will be offered ivabradine alone to allow achievement of targeted heart rate reduction. All patients will be evaluated at 0,6, and 12 months. The end points will be clinical events, cardiac function improvement, renal function, and mortality.

DETAILED DESCRIPTION:
The investigators have already demonstrated the role of targeted heart rate reduction in the management of LVDD in cirrhosis, but the previous study could not demonstrate the role of ivabradine alone in absence of betablocker therapy. This trial will be a validation cohort for the initial data obtained on this novel drug. The use of ivabradine can treat patients who do not tolerate betablocker therapy due to contraindications or adverse effects especially hypotension.

Diagnosis of CCM will be as per 2020 CCMC criteria. CCM is defined as systolic or diastolic dysfunction in the absence of alternative cardiac pathology in concordance with the Cirrhotic Cardiomyopathy Consortium (CCMC) criteria. 9 Systolic dysfunction was defined as an ejection fraction (EF) ≤50% or an absolute value of GLS <18%. CCM will defined as presence of 3 of the following 4 criteria: septal early diastolic mitral annular flow velocity (e') <7 cm/s, early diastolic transmitral flow to early diastolic mitral annular velocity (E/e') ≥15, left atrial volume index (LAVI) >34 mL/m2, tricuspid jet maximum velocity >2.8 m/s, in the absence of pulmonary hypertension and the presence of measurable early to late diastolic transmitral flow velocity (E/A) ratio (E/A >2 = grade 3 & E/A 0.8-2 = grade 2 LVDD). Persons meeting only 2 criteria will be termed as indeterminate for LVDD grade.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-65 years
* Cirrhosis, as diagnosed by histology or clinical, laboratory and USG findings,
* LV diastolic dysfunction on 2D echocardiography

Exclusion Criteria:

* Chronic renal disease
* Patient already on beta blocker
* Pregnancy and peripartum cardiomyopathy
* Hypertension
* Coronary artery disease
* Valvular heart disease
* Sick sinus syndrome/ Pacemaker
* Cardiac rhythm disorder
* Hypothyroidism
* Hyperthyroidism
* Portal vein thrombosis
* Transjugular intrahepatic porto systemic shunt (TIPS) insertion
* Hepatocellular carcinoma
* Anemia Hb < 8gm/dl in females, and < 9 gm/dl in males

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 12 months
  All cause mortality to be assessed

SECONDARY OUTCOMES:
Change in E/e' Ratio | 12 months
  Echo parameter to be documented
Change in renal function | 12 months
Change in HRQoL | 12 months
Change in neurohormonal markers- Brain natriuretic peptide, aldosterone, plasma renin activity | 12 months
Number of Episodes of Cirrhosis related events | 12 months
  New onset ascites, variceal bleeding,hepatorenal syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Radha K Dhiman, MD DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Choose Any State/Province, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Izzy M, VanWagner LB, Lin G, Altieri M, Findlay JY, Oh JK, Watt KD, Lee SS; Cirrhotic Cardiomyopathy Consortium. Redefining Cirrhotic Cardiomyopathy for the Modern Era. Hepatology. 2020 Jan;71(1):334-345. doi: 10.1002/hep.30875. Epub 2019 Oct 11. PMID 31342529
- [Result] Premkumar M, Rangegowda D, Vyas T, Khumuckham JS, Shasthry SM, Thomas SS, Goyal R, Kumar G, Sarin SK. Carvedilol Combined With Ivabradine Improves Left Ventricular Diastolic Dysfunction, Clinical Progression, and Survival in Cirrhosis. J Clin Gastroenterol. 2020 Jul;54(6):561-568. doi: 10.1097/MCG.0000000000001219. PMID 31305281
- [Result] Kaur H, Premkumar M. Diagnosis and Management of Cirrhotic Cardiomyopathy. J Clin Exp Hepatol. 2022 Jan-Feb;12(1):186-199. doi: 10.1016/j.jceh.2021.08.016. Epub 2021 Aug 21. PMID 35068798